CLINICAL TRIAL: NCT06882564
Title: Efficacy of Resveratrol Containing Mouthwash in Reducing Halitosis Related Porphyromonas Gingivalis: A Randomized, Triple-blind Clinical Trial
Brief Title: Efficacy of Resveratrol Containing Mouthwash in Reducing Halitosis Related Porphyrymonas Gingivalis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Nour Ali Abdul, master student, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUOSU-202124
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Halitosis; Mouth Disease; Plaque Induced Gingival Disease; Bleeding Gum; Peridontal Disease
Keywords: halitosis; plaque; gingivitis; resveratrol; chlorhexidine
MeSH Terms: conditions — Halitosis; Mouth Diseases; Gingival Hemorrhage; Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Intervention Model Description: 54 students with halitosis du to gingivitis and interdental plaque accumulation will divided blindly to three groups, each group consisting from 18 patients; The first group will receive anti-oxidant resveratrol mouthwash The second group will receive chlorhexidine mouthwash (positive control group) The third group will receive Distilled water commercially available a placebo mouthwash
Who Masked: Participant, Investigator
Masking Description: the products will be packaged in such a way that they are not recognizable neither by the operator nor by the patient.Each package will be assigned a letter that in turn will refer to the type of product. the association between the letter and the type of product will be collected by another operator .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resveratrol group ( group A ) (Experimental): The participants in this group will receive a resveratrol mouthwash for 7 days, the participants were instructed to rinse twice daily (every 12hours) with 10 ml of the assigned mouthwash (undiluted) for 30 seconds, after 30 minutes of toothbrushing. They will also be provided with measuring cups with 10 ml marking in order to use the correct volume of mouthwash. They were also instructed to refrain from eating and drinking for 30 minutes after rinsing with no change to their routine mechanical dental home care (brushing and interdental aids cleaning). The patients were also informed that burning sensation and bitterness were also expected after rinsing. Discontinuation of the mouthwash was advised in case of any allergic reaction.
  Interventions: Drug: resveratrol mouthwash
- Chlorhexidine group ( group B) (Active Comparator): the participants in this group will receive Chlorhexidine mouthwash for 7 days. they were instructed to rinse twice daily (every 12 hours) with 10 ml of the assigned mouthwash (undiluted) for 30 seconds, after 30 minutes of toothbrushing. They will also be provided with measuring cups with 10 ml markings to use the correct volume of mouthwash. They were also instructed to refrain from eating and drinking for 30 minutes after rinsing with no change to their routine mechanical dental home care (brushing and interdental aid cleaning). The patients were also informed that burning sensations and bitterness were expected after rinsing. Discontinuation of the mouthwash was advised in case of an allergic reaction.
  Interventions: Drug: Chlorhexidine mouthwash (0.2%)
- placebo group ( group C) (Placebo Comparator): the participants in this group will receive a distilled water as amouthwash for 7 days.
  the participants were instructed to rinse twice daily (every 12 hours) with 10 ml of the assigned mouthwash (undiluted) for 30 seconds, after 30 minutes of toothbrushing. They will also be provided with measuring cups with 15 ml markings to use the correct volume of mouthwash. They were also instructed to refrain from eating and drinking for 30 minutes after rinsing with no change to their routine mechanical dental home care (brushing and interdental aid cleaning). The patients were also informed that burning sensations and bitterness were expected after rinsing. Discontinuation of the mouthwash was advised in case of an allergic reaction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: resveratrol mouthwash — the participants where instruct to rinse their mouth twice daily with 10 ml of assigned mouthwash for 60 seconds for 7 days. There is currently no published research on the use of resveratrol as a mouthwash for halitosis treatment.
  This study aims to fill this gap by evaluating its effectiveness in reducing oral malodor through antibacterial action and the potential of volatile sulfur compounds ( VSCs)
  Arms: Resveratrol group ( group A )
Drug: Chlorhexidine mouthwash (0.2%) — The second group will given chlorhexidine 0.2% mouthwash as an active comparator, and will asked to rinse with 10 ml of undiluted mouthwash for 60 seconds twice per day for 7 days, and will instructed to refrain from eating and drinking for 30 min after rinsing.
  Other Names: chlorhexidine 0.2%
  Arms: Chlorhexidine group ( group B)
Drug: Placebo — the third group will given the nonactive control, distilled water, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 seconds twice daily for 7 days and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Other Names: placebo product
  Arms: placebo group ( group C)

SUMMARY:
The aim of the study:

To assess the efficacy of antioxidant (resveratrol) mouthwash in reducing the level of p. gingivitis and oral malodor over 7 day period among undergraduate dental student patients from Mustansiriyah University/College of Dentistry and Wasit University /College of Dentistry.

Objectives:

* To assess the efficacy of anti-oxidant and anti-inflammatory resveratrol mouthwash in reducing halitosis in undergraduate students with plaque-induced gingivitis patients.
* To assess the efficacy of resveratrol mouthwash in reducing p. gingivalis in undergraduate students' patients with oral malodor.
* To determine the relation between p.gingivalis and clinical periodontal parameters (plaque index, gingival index, bleeding on probing) among undergraduate students with plaque-induced gingivitis and halitosis.

DETAILED DESCRIPTION:
54 students with halitosis due to gingivitis and interdental plaque accumulation will divided into three groups, each group consisting of 18 patients; The first group will receive anti-oxidant resveratrol mouthwash The second group will receive chlorhexidine mouthwash (positive control group) The third group will receive Distilled water commercially available as a placebo mouthwash To enhance self-dosing compliance, each participant was contacted each morning and night by text message to remind them to use the mouthwash.

All participants will be subjected to a questionnaire about their name, age, past periodontal treatment, medical history, the medication used, smoking, use of dental brush and interdental aids, and frequency of brushing, the participants will be subjected to another questionnaire about their knowledge, attitude and behaviors about oral malodor, Then (Gingival index, bleeding on probing and plaque index will record clinically All these records will be measured again after one week of using mouthwash twice daily. Finally, the participants filled out a visual analog scale-based assessment questionnaire to obtain feedback on each mouthwash used.

The plaque index will be measured by using the O'Leary plaque index. By recording the presence of plaque on (mesial, distal, facial, lingual) surfaces, A disclosing solution will painted on all exposed tooth surfaces at the initial appointment. The examiner will use an explorer or probe tip to examine all the stained surfaces for dental biofilm. After all teeth were examined and scored, the mean was calculated by dividing the number of plaque surfaces by the total number of available surfaces multiplied by 100%. (O'Leary et al., 1972).

Bleeding on Probing will be measured by gently inserting the periodontal probe at the six surfaces of all teeth to the depth of the gingival sulcus then removing coronally and waiting for 30 seconds to observe the presence or absence of bleeding (0=no bleeding, 1=presence of bleeding). (Newman MG., 2011).

GI will be measured by using Löe and Silness index, each of the four gingival areas of the tooth is given a score from 0 to 3 as follows:

0 Normal gingiva,

1. Mild inflammation slight change in color, slight oedema
2. Moderate inflammation-redness, oedema and glazing.
3. Severe inflammation marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.

the participants will be subjected to organoleptic measurement to detect the patient with halitosis .

The methods used for Organoleptic measurements were done as follows:

1. Tongue odor test: used to determine the halitosis originating from the dorsum of the tongue. A sterile cotton roll was used to scrape the posterior dorsum of the tongue and after 5 seconds the odor is assessed by holding it 5 cm away from the nose (Bosy et al., 1994).
2. Dental floss odor test: used to determine the halitosis originating from the interdental areas. Dental floss pick was passed into the interdental regions of all the teeth by instantly inserting and removing manner and the floss odor is assessed by holding it about 3 cm away from the nose (Ongole and Shenoy, 2010).

A portable sulfide monitor will be use to confirm the result of organoleptic method, a clinical parameter to be measured in logic sequence will include gingival and plaque index. The periodontal examination will be performed by using a periodontal probe.

Randomization and blinding In order to ensure blinding of both participants and the examiner, the mouthwashes will be dispensed into identical opaque bottles measuring 300 ml and each mouthwash group will assign a random sequential letter (A, B, C) and decoding will perform at the end of the study. Microsoft excel (Microsoft Office 2016, Microsoft Corporation, USA) was used to generate random numbers that will be used to resort the order of the mouthwash groups (A, B, C) (N=54) so that each group will receive equal number of participants (N=18) with 1:1:1 allocation. Then, the coded bottles with the mouthwashes were given to the participants together with instructions of use.

All the participants were instructed to rinse twice daily (every 12hours) with 15 ml of the assigned mouthwash (undiluted) for 30 seconds, after 30 minutes of toothbrushing. They will also be provided with measuring cups with 15 ml marking in order to use the correct volume of mouthwash. They were also instructed to refrain from eating and drinking for 30 minutes after rinsing with no change to their routine mechanical dental home care (brushing and interdental aids cleaning). The patients were also informed that burning sensation and bitterness were also expected after rinsing. Discontinuation of the mouthwash was advised in case of any allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* Organoleptic tongue of scores > 2 using (0-5scale) (Rosenberg and McCulloch, 1992)
* Male and female undergraduate dental students without chemical plaque control measures for at least one weak
* Male and female students with halitosis due to gingivitis
* The age of students ranges from 20 to 23 years.
* No periodontal treatment for at least one month
* No systemic disease
* No tobacco smoking
* The patients must have at least 20 teeth

Exclusion Criteria:

* Smokers and alcoholics
* Patient with periodontitis or pocket depth > 6mm
* Patient with orthodontics appliance
* Open carious lesions, pericoronitis, dry socket, and fistula.
* Patients with systemic disease and condition
* taking medication in the last two weeks
* Take garlic, onion, or licorice in the last 24 hours
* using oral hygiene products in the last 24 hours
* pregnant women
* sinusitis, tonsilitis, and upper respiratory tract infection

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
change in oral halitosis (oral malodor) | Baseline (Day 0) and after 7 days
  change in volatile sulfur compounds(VSCs) levels measured by organoleptic method and portable monitor( Halimeter), change in p.gingivalis count using real-time PCR.
  the participants will be subjected to organoleptic measurement to detect the patient with halitosis according to organoleptic categories. A portable sulfide monitor will be use to confirm the result of organoleptic method, a
change in clinical periodontal parameters ( gingival index) | Baseline (Day 0) and after 7 days
  GI will be measured by using Löe and Silness index, each of the four gingival areas of the tooth is given a score from 0 to 3 as follows:
  0 Normal gingiva,
  1. Mild inflammation slight change in color, slight oedema
  2. Moderate inflammation-redness, oedema and glazing.
  3. Severe inflammation marked redness and oedema. Ulceration. Tendency to spontaneous bleeding s
change in clinical periodontal parameters (plaque index) | Baseline (Day 0) and after 7 days
  The plaque index will be measured by using the O'Leary plaque index. By recording the presence of plaque on (mesial, distal, facial, lingual) surfaces, A disclosing solution will painted on all exposed tooth surfaces at the initial appointment. The examiner will use an explorer or probe tip to examine all the stained surface for dental biofilm. After all teeth were examined and scored, the mean was calculated by dividing the number of plaque surfaces by the total number of available surfaces multiplied by 100%. (O'Leary et al., 1972).
change in clinical periodontal parameters (bleeding on probing) | Baseline (Day 0) and after 7 days
  Bleeding on Probing will be measured by gently inserting the periodontal probe at the six surfaces of all teeth to the depth of the gingival sulcus then removed coronally and waited for 30 seconds to observe the presence or absence of bleeding (0=no bleeding, 1=presence of bleeding). (Newman MG., 2011)
change in p.gingivalis level | Baseline (Day 0) and after 7 days
  DNA extraction and purification of p. gingivalis from plaque sample will be performed by using Real-time PCR amplification for each sample using primers specific for p. gingivalis . Bacterial ribosomal RNA (rRNA) primers Will be used to quantify total bacteria both before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: NOOR AA TAHER, B.D.S, Principal Investigator — Al-Mustansiriyah University
Locations (1):
- Mustansiriyah University, Baghdad, Bab Al-Moadham, Iraq

IPD SHARING:
Plan to Share IPD: No
For Privacy concerns, Ethical considerations, Data security and control over data

REFERENCES:
- [Derived] Abed Taher NA, Mahmood AA, Hussein HM. Efficacy of a Mouthwash Containing Resveratrol in Reducing Halitosis-related P. gingivalis: A Randomized Triple-blind Trial. Oral Health Prev Dent. 2025 Dec 2;23:793-803. doi: 10.3290/j.ohpd.c_2373. PMID 41328922